CLINICAL TRIAL: NCT03969966
Title: Citrate Anticoagulation for Postdilution Hemofiltration
Acronym: CIPOHA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Collaborators: Diamed GmbH, Cologne, Germany (Unknown)
Responsible Party: Principal Investigator, Klinik für Anästhesiologie, Prof. Dr. D. Kindgen-Milles, Heinrich-Heine University, Duesseldorf
Other Study IDs: 2018-82
Record Dates: First submitted 2019-05-29; First posted 2019-05-31 (Actual); Last update posted 2020-05-11 (Actual); Status verified 2020-05

CONDITIONS: Acute Kidney Injury; Critical Illness
MeSH Terms: conditions — Acute Kidney Injury; Critical Illness | interventions — Renal Replacement Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: renal replacement therapy as clinically indicated — Continuous renal replacement therapy

SUMMARY:
This study evaluates a protocol for regional citrate anticoagulation in critically ill patients with acute kidney injury who are treated with continuous veno-venous haemofiltration in postdilution mode.

DETAILED DESCRIPTION:
Acute kidney injury (AKI) requiring continuous renal replacement therapy (CCRT occurs in approx. 15 % of all intensive care patients. A sustained and prolonged filter running time is required to deliver an effective dialysis dose. This requires effective anticoagulation. Today, regional citrate anticoagulation (RCA) is preferred over systemic anticoagulation because of prolonged filter lifetimes and less adverse effects.

We here study prospectively patients with AKI who are treated with continuous veno-venous haemofiltration using an RCA protocol.

We will evaluate all parameters of CRRT including filter running times, delivered dialysis dose, causes for treatment interruption and control of pH and electrolytes.

ELIGIBILITY:
Inclusion Criteria:

* acute kidney injury
* critical illness and treatment at ICU

Exclusion Criteria:

* age < 18 years
* pregnancy or breast feeding
* severe lactate acidosis ( > 10 mmol/l) for longer than 6 hours and pH < 7.2

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Critically ill patients at ICU with acute kidney injury
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-01-14 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
Filter running time | 72 hours
  Filterlifetime with regional citrate anticoagulation for haemofiltration

CONTACTS AND LOCATIONS:
Locations (1):
- Intensivstation ZOM1 Klinik für Anästhesiologie Universitätsklinikum Düsseldorf, Düsseldorf, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Dimski T, Brandenburger T, Vollmer C, Kindgen-Milles D. A safe and effective protocol for postdilution hemofiltration with regional citrate anticoagulation. BMC Nephrol. 2024 Jul 9;25(1):218. doi: 10.1186/s12882-024-03659-y. PMID 38982339